CLINICAL TRIAL: NCT07115082
Title: A Randomized, Open-label, Parallel-controlled Clinical Study of Amniotic Mesenchymal Stem Cells in the Treatment of Premature Ovarian Insufficiency
Brief Title: Clinical Study on the Safety and Efficacy of Human Amniotic Mesenchymal Stem Cells in the Treatment of Premature Ovarian Insufficiency
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yan Hongli (Other)
Responsible Party: Sponsor-Investigator, Yan Hongli, Professor of Reproductive Medicine, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHEC2023-172
Record Dates: First submitted 2025-03-26; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Premature Ovarian Insufficiency
Keywords: hA-MSCs; Premature ovarian insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Climen (Active Comparator): Hormone replacement therapy (HRT): Take the drug Climen. Each box has 21 tablets. The first 11 tablets contain 2 milligrams of estradiol valerate each. The last 10 tablets contain 2 milligrams of estradiol valerate and 1 milligram of cyproterone acetate each. Begin taking it on the fifth day of your menstrual cycle. Take one tablet every day for seven days. Then, stop taking the medicine for seven days. After that, continue for two cycles in a row.
  Interventions: Drug: Climen 21 Tablets
- hA-MSCs+Climen (Experimental): The stem cell treatment group will be administered Climen, with the dosage and method of administration to be determined based on the control group. Concurrently, patients will receive the initial infusion of amniotic MSCs intravenously on the third day after the onset of menstruation, with a subsequent infusion administered after one month. The number of stem cells infused was calculated according to 1 million cells per kilogram of body weight.
  Interventions: Drug: Climen 21 Tablets; Biological: hA-MSCs

INTERVENTIONS:
Drug: Climen 21 Tablets — Climen is commonly used clinically as a hormone replacement therapy and was administered to all patients in both the control and experimental groups in this project.
Biological: hA-MSCs — The patients who were part of the experimental group were administered oral Clomid medication in conjunction with a combined intravenous injection of human amniotic MSCs.
  Arms: hA-MSCs+Climen

SUMMARY:
There is a high incidence of women suffering from Primary Ovarian Insufficiency (POI). So far, there was no treatment sufficient enough to cure POI. Cell therapy is a rapidly developing field and have shown immense promise in the treatment of ovarian dysfunction. In this study, the investigator will evaluate the safety of human Amniotic mesenchymal stem cells (hA-MSCs) therapy in women suffering from POI.

DETAILED DESCRIPTION:
This clinical trial is designed to understand the safety and effectiveness of human amniotic membrane mesenchymal stem cells (hA-MSCs) in the treatment of primary ovarian insufficiency (POI). Human amniotic MSCs were infused back into the patients by intravenous injection. The trial was designed with two groups, 1) the control group by conventional hormone replacement therapy with oral Climen and 2) the stem cell treatment group by intravenous infusion of human amniotic membrane mesenchymal stem cells (hA-MSCs) combined with oral Climen hormone therapy. Patients were followed up every 2 weeks after the post-injection stem cells to observe their outcomes. The investigators focused on safety indicators, but also monitored hormone levels and signs of follicular growth to initially assess the effectiveness of the stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. The intention of pregnant women aged >= 20 and < 40, with normal karyotype;
2. Oligo/amenorrhea for at least 4 months;
3. Elevated FSH level >25 IU/l on two occasions >4 weeks apart;
4. Without a history of stem cell therapy and no growth hormone and/or estrogen and progesterone therapy within the previous 3 months;
5. Voluntary participation in the study with signed informed consent;

Exclusion Criteria:

1. Unable to follow the treatment observation process required by the trial;
2. Genetic diseases, chromosomal abnormalities, and genetic deficiency that clearly cause premature ovarian insufficiency/premature ovarian failure;
3. With breast, uterine, ovarian tumors, or any other benign or malignant tumors;
4. Allergic history to drugs or any other things;
5. Presence of genetic disorders such as Turner's syndrome, congenital malformations of the reproductive organs.
6. Have undergone ovariectomy or have organic gynaecological diseases.
7. Presence of other gynaecological endocrine diseases such as polycystic ovary syndrome.
8. Severe functional impairment of vital organs.
9. High risk factors for venous thromboembolism and abnormalities in coagulation mechanisms.
10. Attending doctor considers inappropriate to take part in.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Temperature | Up to 24 weeks
  Body temperature of the participants will be measured fortnightly after injection.
Pulse | up to 24 weeks
  Pulse of the participants will be measured fortnightly after injection.
Breaths per minute | up to 24 weeks
  Breathing rate of the participants will be measured fortnightly after injection.
Blood pressure | 0-24 weeks
  Both systolic pressure and diastolic pressure of the participants will be assessed fortnightly after injection.

SECONDARY OUTCOMES:
Follicle-stimulating hormone (FSH) serum level | Up to 24 weeks
  Serum FSH level will be tested fortnightly after injection.
Estradiol (E2) serum level | Up to 24 weeks
  Serum E2 level will be tested fortnightly after injection.
Anti-Mullerian hormone (AMH) serum level | up to 24 weeks
  Serum AMH level will be tested fortnightly after injection.
Number of antral follicle | up to 24 weeks
  The number of antral follicles developing will be recorded by transvaginal ultrasound fortnightly after injection.
Achievement of pregnancy | up to 12 months
  A transvaginal ultrasound confirmation of gestational sac The hCG levels have reached between 1,000 - 2,000 mIU/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided